CLINICAL TRIAL: NCT01118624
Title: Phase 2 Study of Pralatrexate in Female Patients With Previously-treated Advanced or Metastatic Breast Cancer
Brief Title: Study of Pralatrexate in Female Patients With Previously-treated Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-014; 2008-006425-14 (EudraCT Number)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Breast Tumors; Neoplasms, Breast; Cancer of the Breast; Human Mammary Carcinoma
Keywords: Female; Advanced; Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — 10-propargyl-10-deazaaminopterin; Vitamin B 12; Folic Acid

ARMS (1):
- Pralatrexate, (RS)-10-propargyl-10-deazaaminopterin (Folotyn) (Experimental): Intravenous (IV) push administration over 3-5 minutes. Initial dose: 190 mg/m2 Dose reductions per protocol: 150 mg/m2, 120 mg/m2, and 100 mg/m2 allowed for defined toxicities.
  Administered on days 1 and 15 of a 4-week cycle (every 2 weeks) until criteria for discontinuation per the protocol are met.
  Interventions: Drug: Pralatrexate Injection; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Pralatrexate Injection — Intravenous (IV) push administration over 3-5 minutes.
  Initial dose: 190 mg/m2
  Dose reductions per protocol: 150 mg/m2, 120 mg/m2, and 100 mg/m2 allowed for defined toxicities.
  Administered on days 1 and 15 of a 4-week cycle (every 2 weeks) until criteria for discontinuation per the protocol are met.
  Other Names: FOLOTYN; Pralatrexate; PDX; (RS)-10-propargyl-10-deazaaminopterin
Dietary Supplement: Vitamin B12 — 1 mg intramuscular injection
  Administered within 10 weeks prior to first dose of pralatrexate, every 8-10 weeks throughout the study and for at least 30 days after the last dose of pralatrexate.
  Other Names: Cyanocobalamin
Dietary Supplement: Folic Acid — 1.0-1.25 mg orally
  Administered daily for at least 7 days prior to first dose of pralatrexate, throughout the study and for at least 30 days after the last dose of pralatrexate.
  Other Names: Vitamin B9; Folate; Folacin

SUMMARY:
The purpose of this study is to determine the efficacy (ability to provide a beneficial treatment of the disease) of pralatrexate for the treatment of female patients with advanced or metastatic breast cancer who have failed prior chemotherapy. Patients will receive vitamin B12 and folic acid supplementation.

DETAILED DESCRIPTION:
This is an open label, multi-center, Phase 2 study of pralatrexate with vitamin B12 and folic acid supplementation in patients with advanced or metastatic breast cancer who have failed prior treatment(s).

The start of study treatment is defined as the initiation of pralatrexate administration.

Pralatrexate will be administered as an intravenous (IV) push over 3-5 minutes on days 1 and 15 (± 1 day at each time point) of a 4-week cycle (ie, every [q] 2 weeks). The initial dose of pralatrexate will be 190 mg/m2. Dose reduction to 150 mg/m2 with further reduction to 120 mg/m2 and 100 mg/m2 will be allowed for defined toxicity (see Section 7.3). If 100 mg/m2 is not tolerated, pralatrexate must be discontinued.

Patients will receive vitamin supplementation consisting of vitamin B12, 1 mg intramuscular (IM) q 8-10 weeks and folic acid 1-1.25 mg by mouth (PO) once a day (QD). Patients must have received 1 mg vitamin B12 within 10 weeks prior to the initiation of pralatrexate and have received 7 days of 1-1.25 mg folic acid PO QD prior to the initiation of pralatrexate.

Vitamin supplementation will continue throughout the study and for at least 30 days after the last administration of pralatrexate.

ELIGIBILITY:
Inclusion Criteria:

* HER-2 negative advanced or metastatic breast cancer
* Disease has become worse after at least 1 prior chemotherapy regimen for advanced or metastatic disease
* Advanced or metastatic disease resistant to both a taxane and an anthracycline-containing chemotherapy regimen, or resistant to taxanes and for whom further anthracycline therapy is not indicated
* Patients with controlled brain metastases must have finished receiving radiation therapy and if on corticosteroids, be on a stable or tapering dose of ≤ 10 mg/day of prednisone or equivalent for at least 28 days prior to study entry
* Measurable disease
* Female 18 years of age or older
* Performance status less than or equal to 2
* Life expectancy of more than 3 months
* Blood, liver and kidney laboratory test results that meet protocol requirements
* Patients must have a negative serum pregnancy test within 14 days before enrollment and agree to use medically acceptable and effective birth control from enrollment until at least 30 days after the last dose of pralatrexate. Patients who are postmenopausal for at least 1 year (more than 12 months since last menses) or are surgically sterilized do not require this test.
* Willing to attend visits for repeat dosing and follow up
* Give written informed consent

Exclusion Criteria:

* Patients with only bone metastasis
* Patients with a single metastatic site without histological proof that the lesion is metastatic breast cancer
* Patients with inflammatory breast cancer
* Treatment with systemic chemotherapy, hormone therapy, radiation therapy, or other investigational therapy within 3 weeks (6 weeks for nitrosoureas, mitomycin C) prior to enrollment, except for the following:

  * Bisphosphonates, if ongoing
  * Prior treatment with methotrexate
  * Prior treatment with anti-angiogenics within 6 months prior to enrollment
* Have received more than 2 prior chemotherapy regimens (more than 3 if one of the treatments was neoadjuvant or adjuvant chemotherapy)
* Have previously received pralatrexate
* Have received more than the allowed maximum total dose of anthracycline
* Prior radiation therapy on more than 30% of bone marrow reserve or prior bone marrow/stem cell transplantation
* Congestive heart failure Class III/IV
* Uncontrolled hypertension (high blood pressure)
* Active infection or any serious medical condition, which would impair the ability of the patient to receive protocol treatment
* Females who are pregnant or breastfeeding
* Major surgery within 14 days of enrollment
* Another active cancer in addition to advanced or metastatic breast cancer, except well treated in situ cervical cancer and basal cell skin cancer
* Dementia or other altered mental status that would prevent the patient from understanding and giving informed consent or limit her ability to follow the study requirements
* Patients who are human immunodeficiency virus (HIV)-positive and have a CD4 count of less than 100 mm3 or detectable viral load within past 3 months and is receiving anti-retroviral therapy
* Patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) who have a detectable viral load or immunological evidence of chronic active disease or receiving/requiring antiviral therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garry Weems, PharmD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (14):
- United States (2):
  - Providence Cancer Center, Portland, Oregon
  - The West Clinic, Memphis, Tennessee
- Czechia (3):
  - Fakultní nemocnice Olomouc, Olomouc
  - Multiscan, s.r.o., Pardubice
  - Fakultní nemocnice Královské Vinohrady - FNKV, Prague
- France (6):
  - Centre Lutte Contre le Cancer Val d'Aurelle (CRLC), Montpellier, Cedex 5
  - Centre Régional de Lutte Contre le Cancer Alexis Vautrin, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Jean-Godinot, Reims
- Hungary (3):
  - University of Debrecen Medical and Health Science Center, Debrecen, Hajdú-Bihar
  - Semmelweis University Budapest, Budapest
  - National Health Centre of Hungary, Budapest

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 05 Oct 2009 and 10 May 2011. Patients were enrolled in Hungary, France, and the Czech Republic.
Groups:
- Pralatrexate: Study drug 190 mg/m^2 for 2 to 4 weeks.
Period: Overall Study
Arm/Group | Pralatrexate
Started | 22
Completed | 0
Not Completed | 22

BASELINE CHARACTERISTICS:
Population: Patients enrolled and treated with study drug.
Arm/Group | Pralatrexate
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Tumor response evaluation was performed using RECIST 1.0 using CT/MRI. Proportion of patients achieving a CR or PR is considered in the overall response.
Time Frame: Assessed at the end of each even-numbered cycle (every 8 weeks), or per standard of care but no less than 4 weeks and nor more than every 12 weeks (+/- 1 week) if treatment has ended.
Measure: Number; unit: participants
Arm/Group | Pralatrexate
Number analyzed (Participants) | 22
participants | 1 [0.1 to 22.8]

2. Secondary Outcome: Duration of Response (DOR)
Description: One patient has a PR as response and duration of response was provided for that patient.
Time Frame: as for outcome 1
Measure: Number; unit: days
Arm/Group | Pralatrexate
Number analyzed (Participants) | 1
days | 112

3. Secondary Outcome: Overall Survival (OS)
Description: Number of days from first dose of pralatrexate to death.
Time Frame: Assessed at the end of each even-numbered cycle (every 8 weeks), or per standard of care but at least every 4 weeks and no more than every 12 weeks (+/- 1 week) if treatment has ended. OS will be collected for up to 2 years from start of pralatrexate.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 22
months | 11.3 [6.8 to 13.9]

4. Secondary Outcome: Incidence of Adverse Events (AEs) and Laboratory Abnormalities
Time Frame: Recorded at all study visits: every 2 weeks while on treatment and at safety follow-up (35 +/- 5 days post-last dose) or early termination visit (at time of withdrawal).
Measure: Number; unit: participants
Arm/Group | Pralatrexate
Number analyzed (Participants) | 22
participants | 21

ADVERSE EVENTS:
Time Frame: All treated patients will be followed for safety through 35 (± 5) days after their last dose or until all treatment-related AEs have resolved or returned to baseline/Grade 1, whichever is longer
Arm/Group | Pralatrexate
Serious Adverse Events (participants affected / at risk) | 6/22
Other Adverse Events (participants affected / at risk) | 1/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralatrexate (N=22)
MUCOSAL INFLAMMATION (Gastrointestinal disorders) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pralatrexate (N=22)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Sufficient patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No